CLINICAL TRIAL: NCT00157313
Title: Randomised Clinical Trial of Integrated Treatment Versus Standard Treatment in First Episode Psychosis
Brief Title: Clinical Trial of Integrated Treatment Versus Standard Treatment in First Episode Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); Ministry of Social Affairs, Denmark (Other Government); University of Copenhagen (Other); Copenhagen Hospital Corporation (Other); Medical Research Council (Other Government); Wørzners Foundation. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPUS trial
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2005-09

CONDITIONS: Psychotic Disorders; Schizophreniform Disorders; Schizoaffective Disorder; Psychosis, Brief Reactive; Schizophrenia, Borderline
Keywords: Schizophrenia; First episode psychosis; Psychosocial intervention
MeSH Terms: conditions — Psychotic Disorders; Schizotypal Personality Disorder; Schizophrenia

INTERVENTIONS:
Behavioral: Integrated treatment, family involvement
Behavioral: Social skills training

SUMMARY:
The purpose of the study was to evaluate the effects of integrated treatment for patients with a first episode of psychotic illness. We conducted a randomised clinical trial in Copenhagen Hospital Corporation and Psychiatric Hospital Aarhus, Denmark. We included 547 patients with first episode of schizophrenia spectrum disorder, who has not received antipsychotic medication for more than 12 weeks.

Patients were randomised to integrated treatment or standard treatment. The integrated treatment lasted for two years and consisted of assertive community treatment with programmes for family involvement and social skills training. Standard treatment offered contact with a community mental health centre.

We wanted to study the effect on psychotic (hallucinations and delusions)and negative (lack of initiative, apati, blunted affect) symptoms (each scored from 0 to a maximum of 5) at one and two years' follow-up.

We found that integrated treatment improved clinical outcome and adherence to treatment. The improvement in clinical outcome was consistent at one year and two year follow-ups. We will study further outcome measures such as social network, quality of life, depression and suicidal behaviour.

DETAILED DESCRIPTION:
Objectives: To evaluate the effects of integrated treatment for patients with a first episode of psychotic illness.

Design: Randomised clinical trial. Setting: Copenhagen Hospital Corporation and Psychiatric Hospital Aarhus, Denmark Participants: 547 patients with first episode of schizophrenia spectrum disorder.

Interventions: Integrated treatment and standard treatment. The integrated treatment lasted for two years and consisted of assertive community treatment with programmes for family involvement and social skills training. Standard treatment offered contact with a community mental health centre.

Main outcome measures: Psychotic and negative symptoms (each scored from 0 to a maximum of 5) at one and two years' follow-up.

Results: At one year's follow-up, psychotic symptoms changed favourably to a mean of 1.09 (standard deviation 1.27) with an estimated mean difference between groups of -0.31 (95% confidence interval -0.55 to -0.07, P=0.02) in favour of integrated treatment. Negative symptoms changed favourably with a estimated difference between groups of -0.36 (-0.54 to -0.17, P<0.001) in favour of integrated treatment. At two years' follow-up the estimated mean difference between groups in psychotic symptoms was -0.32 (-0.58 to -0.06, P=0.02) and in negative symptoms was -0.45 (-0.67 to -0.22, P<0.001), both in favour of integrated treatment. Patients who received integrated treatment had significantly less comorbid substance misuse, better adherence to treatment, and more satisfaction with treatment.

Conclusion: Integrated treatment improved clinical outcome and adherence to treatment. The improvement in clinical outcome was consistent at one year and two year follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* F2 diagnosis in ICD 10
* Address in Copenhagen, Frederiksberg or Aarhus
* Antipsychotic medication not exceeding 12 weeks
* Informed consent

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600
Dates: Start 1998-01; Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Psychotic symptoms at one and two year follow-up
Negative symptoms at one and two year follow-up

SECONDARY OUTCOMES:
Adherence at one and two year follow-up
Depression at one and two year follow-up
Suicidal behaviour at one and two year follow-up
Use satisfaction at one and two year follow-up
Quality of life at one and two year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Ph.D., Principal Investigator — Bispebjerg Hospital, department of psychiatry, University of Copenhagen
Locations (1):
- Bispebjerg Hospital, department of psychiatry, Copenhagen, Denmark

REFERENCES:
- [Background] Jorgensen P, Nordentoft M, Abel MB, Gouliaev G, Jeppesen P, Kassow P. Early detection and assertive community treatment of young psychotics: the Opus Study Rationale and design of the trial. Soc Psychiatry Psychiatr Epidemiol. 2000 Jul;35(7):283-7. doi: 10.1007/s001270050240. PMID 11016522
- [Result] Nordentoft M, Jeppesen P, Abel M, Kassow P, Petersen L, Thorup A, Krarup G, Hemmingsen R, Jorgensen P. OPUS study: suicidal behaviour, suicidal ideation and hopelessness among patients with first-episode psychosis. One-year follow-up of a randomised controlled trial. Br J Psychiatry Suppl. 2002 Sep;43:s98-106. doi: 10.1192/bjp.181.43.s98. PMID 12271808
- [Result] Petersen L, Jeppesen P, Thorup A, Abel MB, Ohlenschlaeger J, Christensen TO, Krarup G, Jorgensen P, Nordentoft M. A randomised multicentre trial of integrated versus standard treatment for patients with a first episode of psychotic illness. BMJ. 2005 Sep 17;331(7517):602. doi: 10.1136/bmj.38565.415000.E01. Epub 2005 Sep 2. PMID 16141449
- [Result] Thorup A, Petersen L, Jeppesen P, Ohlenschlaeger J, Christensen T, Krarup G, Jorgensen P, Nordentoft M. Integrated treatment ameliorates negative symptoms in first episode psychosis--results from the Danish OPUS trial. Schizophr Res. 2005 Nov 1;79(1):95-105. doi: 10.1016/j.schres.2004.12.020. PMID 16122909
- [Result] Petersen L, Nordentoft M, Jeppesen P, Ohlenschaeger J, Thorup A, Christensen TO, Krarup G, Dahlstrom J, Haastrup B, Jorgensen P. Improving 1-year outcome in first-episode psychosis: OPUS trial. Br J Psychiatry Suppl. 2005 Aug;48:s98-103. doi: 10.1192/bjp.187.48.s98. PMID 16055817
- [Result] Jeppesen P, Petersen L, Thorup A, Abel MB, Oehlenschlaeger J, Christensen TO, Krarup G, Hemmingsen R, Jorgensen P, Nordentoft M. Integrated treatment of first-episode psychosis: effect of treatment on family burden: OPUS trial. Br J Psychiatry Suppl. 2005 Aug;48:s85-90. doi: 10.1192/bjp.187.48.s85. PMID 16055815
- [Result] Rosenbaum B, Valbak K, Harder S, Knudsen P, Koster A, Lajer M, Lindhardt A, Winther G, Petersen L, Jorgensen P, Nordentoft M, Andreasen AH. The Danish National Schizophrenia Project: prospective, comparative longitudinal treatment study of first-episode psychosis. Br J Psychiatry. 2005 May;186:394-9. doi: 10.1192/bjp.186.5.394. PMID 15863743
- [Derived] Starzer MSK, Hansen HG, Hjorthoj C, Speyer H, Albert N, Nordentoft M. Predictors of Mortality Following a Schizophrenia Spectrum Diagnosis: Evidence From the 20-Year Follow-up of the OPUS Randomized Controlled Trial. Schizophr Bull. 2023 Sep 7;49(5):1256-1268. doi: 10.1093/schbul/sbad111. PMID 37527479
- [Derived] Hansen HG, Starzer M, Nilsson SF, Hjorthoj C, Albert N, Nordentoft M. Clinical Recovery and Long-Term Association of Specialized Early Intervention Services vs Treatment as Usual Among Individuals With First-Episode Schizophrenia Spectrum Disorder: 20-Year Follow-up of the OPUS Trial. JAMA Psychiatry. 2023 Apr 1;80(4):371-379. doi: 10.1001/jamapsychiatry.2022.5164. PMID 36811902
- [Derived] Madsen T, Karstoft KI, Secher RG, Austin SF, Nordentoft M. Trajectories of suicidal ideation in patients with first-episode psychosis: secondary analysis of data from the OPUS trial. Lancet Psychiatry. 2016 May;3(5):443-50. doi: 10.1016/S2215-0366(15)00518-0. Epub 2016 Mar 3. PMID 26948484
- [Derived] Jeppesen P, Petersen L, Thorup A, Abel MB, Ohlenschlaeger J, Christensen TO, Krarup G, Jorgensen P, Nordentoft M. The association between pre-morbid adjustment, duration of untreated psychosis and outcome in first-episode psychosis. Psychol Med. 2008 Aug;38(8):1157-66. doi: 10.1017/S0033291708003449. Epub 2008 Apr 30. PMID 18447961